CLINICAL TRIAL: NCT06090058
Title: Role of Neurofilament Light Chain as a Diagnostic Tool and Predictor of Outcome of Acute Ischemic Stroke.
Brief Title: NF-L Chain Measurement in Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolous Hana Henein, Resident, Assiut University
Other Study IDs: NF-L chain in acute stroke
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: Patients with acute ischemic stroke having focal neurological deficits lasting for more than 24 hour with relevant lesion in brain computerized tomography (CT) or magnetic resonance (MR) image
  Interventions: Diagnostic Test: Measurement of neurofilament light chain
- B: Patients with chronic ischemic stroke , having these symptoms for 6-12 month
  Interventions: Diagnostic Test: Measurement of neurofilament light chain
- C: Healthy controls
  Interventions: Diagnostic Test: Measurement of neurofilament light chain

INTERVENTIONS:
Diagnostic Test: Measurement of neurofilament light chain — Serum samples will be collected into a serum gel with clotting activator tube (Sarstedt). After delivery to the laboratory, the serum samples were centrifuged at 2500 × g for 6 min at 4 Celsius degree, then aliquoted into at least three vials (0.3 mL per vial) and stored at -70 Celsius degree until the analysis.

SUMMARY:
1. Using neurofilament light chain as a diagnostic tool and predictor of outcome of acute ischemic stroke
2. Using neurofilament light chain in detecting severity in old ischemic stroke

DETAILED DESCRIPTION:
Ischemic stroke is the second leading cause of death and disability with symptoms ranging from complete remission within 24 h (transient ischemic attack, TIA) to lasting disability in the form of cognitive dysfunction, physical disability, and complete dependency on others. The currently available acute treatments of intravenous administration of tissue plasminogen activator (2) and mechanical thrombectomy are associated with rare but severe side effects such as hemorrhage of the brain and body. Because these treatments require rapid initiation to be effective, some patients may be exposed to side effects without benefiting from the treatment. We need, therefore, to identify biomarkers that can predict functional outcome, especially in the early phases, and improve our understanding of the pathophysiological mechanisms underlying tissue damage following a stroke to develop new advanced therapeutic strategies.

When brain damage occurs, neuronal injury and disruption of axonal membranes lead to the release of cytoskeleton proteins, such as neurofilaments (NFs), into the interstitial fluid and eventually into the cerebrospinal fluid (CSF) and blood. NFs are highly specific structural, neuronal cytoskeletal proteins that consist of four NF subunits: NF light (NF-L), NF medium (NFM), and NF heavy (NF-H) chains, and alpha-internexin.

NF-L has been studied as a potential CSF and circulation biomarker for a wide range of neurological disorders (3), including cerebral small vessel disease (4) and subacute ischemic stroke.

The inflammatory process that ensues after a stroke destabilizes the blood-brain barrier (BBB) and contributes to neuro-axonal damage, thereby increasing the release of NFs and glial and inflammatory markers into the CSF and blood.

Ischemic stroke has recently been shown to cause persistent elevations in serum NF-L that correlated with infarct volumes and recurrent ischemic lesions.

So, Measuring serum level of NF-L will be promising as a biomarker for predicting severity of stroke symptoms and its functional outcome. So, we can predict prognosis of these cases.

NF-L levels obtained within 24 h of symptom onset in the blood of ischemic stroke and TIA patients will be associated with diagnosis of these patients and as a predictor for functional outcome of these patients.

These patients after 1 and 3 months will be assessed again clinically by NIHSS and mRS to assess their outcome and detecting possibility of recurrence.

the investigators will also measure serum NF-L levels in old ischemic stroke patients having stroke of 6 to 12 month duration, as NF-L will be used as a predictor of severity of ischemic stroke in these patients.

the investigators will also measure NF-L in healthy controls to compare its level between the healthy and diseased cases.

the investigators will also measure infarct size in MR imaging, measure media-intima thickness of carotid artery, and correlate their findings with NF-L serum level to predict stroke severity and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* both sex
* Age between 18 to 70 years old.
* symptoms suggestive of acute ischemic stroke: presenting within 24 hours of onset of these symptoms
* for chronic ischemic patients : Duration of 6 to 12 month of development of ischemic symptoms
* for control cases : Healthy people

Exclusion Criteria:

* presence of space occupying lesion
* presence of sinus thrombosis
* presence of hemorrhagic stroke
* presence of sub-arachnoid hemorrhage
* presence of Alzheimer disease, Parkinson disease, multiple sclerosis, amyotrophic lateral sclerosis, or traumatic brain injury

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: population will include 3 groups, group A : will include patients of acute ischemic stroke - developing focal neurological symptoms in first 24 hour - of age between 18 - 70 year old.
  group B : will include patients of chronic ischemic stroke - developing focal neurological symptoms for 6-12 month - of age between 18 - 70 year old. group C : will be healthy controls of age above 18 y.o
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
measuring neurofilament light chain in stroke patients | baseline
  correlation between levels of neurofilament light chain with severity and functional outcome of stroke patients

REFERENCES:
- [Background] Ahn JW, Hwang J, Lee M, Kim JH, Cho HJ, Lee HW, Eun MY. Serum neurofilament light chain levels are correlated with the infarct volume in patients with acute ischemic stroke. Medicine (Baltimore). 2022 Sep 30;101(39):e30849. doi: 10.1097/MD.0000000000030849. PMID 36181119
- [Background] Banks JL, Marotta CA. Outcomes validity and reliability of the modified Rankin scale: implications for stroke clinical trials: a literature review and synthesis. Stroke. 2007 Mar;38(3):1091-6. doi: 10.1161/01.STR.0000258355.23810.c6. Epub 2007 Feb 1. PMID 17272767
- [Background] Revendova KZ, Zeman D, Bunganic R, Karasova K, Volny O, Bar M, Kusnierova P. Serum neurofilament levels in patients with multiple sclerosis: A comparison of SIMOA and high sensitivity ELISA assays and contributing factors to ELISA levels. Mult Scler Relat Disord. 2022 Nov;67:104177. doi: 10.1016/j.msard.2022.104177. Epub 2022 Sep 11. PMID 36130459
- [Background] Gaiottino J, Norgren N, Dobson R, Topping J, Nissim A, Malaspina A, Bestwick JP, Monsch AU, Regeniter A, Lindberg RL, Kappos L, Leppert D, Petzold A, Giovannoni G, Kuhle J. Increased neurofilament light chain blood levels in neurodegenerative neurological diseases. PLoS One. 2013 Sep 20;8(9):e75091. doi: 10.1371/journal.pone.0075091. eCollection 2013. PMID 24073237
- [Background] Nielsen HH, Soares CB, Hogedal SS, Madsen JS, Hansen RB, Christensen AA, Madsen C, Clausen BH, Frich LH, Degn M, Sibbersen C, Lambertsen KL. Acute Neurofilament Light Chain Plasma Levels Correlate With Stroke Severity and Clinical Outcome in Ischemic Stroke Patients. Front Neurol. 2020 Jun 11;11:448. doi: 10.3389/fneur.2020.00448. eCollection 2020. PMID 32595585